CLINICAL TRIAL: NCT01687660
Title: A Continuous Study on Abiding Effect of Acupuncture for Migraine Treatment
Brief Title: Acupuncture for Migraine Prophylaxis
Acronym: AMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Li ying (Other)
Collaborators: Hunan University of Traditional Chinese Medicine (Other); Chongqing Medical University (Other)
Responsible Party: Sponsor-Investigator, Li ying, Chengdu University of Traditional Chinese Medicine, Chengdu University of Traditional Chinese Medicine
Organization: Chengdu University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012CB518501-2
Record Dates: First submitted 2012-08-31; First posted 2012-09-19 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Migraine Without Aura; Unilateral Headache
Keywords: acupuncture; migraine prophylaxis
MeSH Terms: conditions — Migraine without Aura; Headache | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- acupoint-meridian group (Experimental): Apply traditional acupuncture to prevent the migraine attack according to TCM theory
  Interventions: Other: acupuncture
- sham-acupoint group (Other): sham-acupoint will be penetrated for migraine prophylaxis.
  Interventions: Other: acupuncture
- waiting list (No Intervention): No acupuncture nor other methods will be conducted in this group.

INTERVENTIONS:
Other: acupuncture — apply acupuncture to prevent the migraine attack
  Arms: acupoint-meridian group; sham-acupoint group

SUMMARY:
Hypothesis: Acupuncture obtains an abiding effect on migraine prophylaxis Design: A open-label randomized controlled trial. 249 participants will be included. Three arms: acupuncture in acupoint-meridian， non-acupoint-meridian group, and waiting list.

DETAILED DESCRIPTION:
Aim: to attest the abiding efficacy and safety of acupuncture for migraine prophylaxis Design: A open-label randomized controlled trial will be performed in Chengdu, Hunan and Chongqing province. Two hundred and forty-three participants will be randomly assign to acupoint-meridian group, non-acupoint-meridian group, and wait-and-see group. Each participants will receive 20 sessions of acupuncture in 4 weeks, with a duration of 30 minutes in a session. After all the treatments was accomplished, there will be 5 times follow-ups in the impending every 4 weeks. The primary outcome is frequency of migraine attacks 16 weeks after inclusion. Secondary outcomes include frequency of migraine attacks at the 4th and 24th week, headache severity, MSQ(Migraine Specific Quality of Life Questionnaire MSQ Version2.1), etc.

ELIGIBILITY:
Inclusion Criteria:

* Age of a subject is between 18 and 65 years old(initially occured beneath the age of 50), male or female;
* in accordance with diagnosis of migraine without aura in International Classification of Headache Disorders, ICHD-2, by IHS;
* 2 to 8 times attack per month in recent 3 months, with each period beyond 15 days;
* with migraine history for over 1 year;
* be able and willing to finish the headache diary in baseline ;
* informed consent form must be signed by patient or lineal relative;

Exclusion Criteria：

* Patients who are unconscious, psychotic.
* Patients with aggravating tumor and other serious consumptive disease, and who are subject to infection and bleeding.
* With serious primary illness or disease of cardiovascular, liver, renal, gastrointestinal, hematological systems and so on.
* Pregnant women or women in lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
frequency of migraine attacks | 16th week after inclusion
  to assess the frequency of migraine attacks at the 16th week after inclusion

SECONDARY OUTCOMES:
frequency of migraine attacks | 4th and 24th week after inclusion
  to assess the frequency of migraine attacks at the 4th and 24th week respectively
headache severity | 0 day, 4th, 8th, 12th, 16th, 20th, 24th week after inclusion
  to evaluate the change of severity of headache

OTHER OUTCOMES:
MSQ(Migraine Specific Quality of Life Questionnaire MSQ Version2.1) | the day of inclusion and 4th week after inclusion
  to observe the change of MSQ
acupuncture expectation scale | 1 day
  an outcome to indicate the expectation of patient towards acupuncture treatment for migraine

CONTACTS AND LOCATIONS:
Overall Officials: Fanrong Liang, Professor, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu University of TCM, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhao L, Chen J, Li Y, Sun X, Chang X, Zheng H, Gong B, Huang Y, Yang M, Wu X, Li X, Liang F. The Long-term Effect of Acupuncture for Migraine Prophylaxis: A Randomized Clinical Trial. JAMA Intern Med. 2017 Apr 1;177(4):508-515. doi: 10.1001/jamainternmed.2016.9378. PMID 28241154
- [Derived] Chen J, Zhao L, Zheng H, Li Y, Yang M, Chang X, Gong B, Huang Y, Liu Y, Liang F. Evaluating the prophylaxis and long-term effectiveness of acupuncture for migraine without aura: study protocol for a randomized controlled trial. Trials. 2013 Oct 30;14:361. doi: 10.1186/1745-6215-14-361. PMID 24171782